CLINICAL TRIAL: NCT04577885
Title: A Single-center, Open, Single Does, Drug-drug Interaction Study to Investigate the Effects of Rifampin on the Pharmacokinetics of Healthy Chinese Adult Subjects After Oral Administration of SHR2554 Tablets
Brief Title: A Rifampin Effect Study of SHR2554 on Healthy Chinese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHR2554-I-107
Record Dates: First submitted 2020-09-24; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Healthy
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Single-dose oral administration of SHR2554 and multiple-dose oral administration of Rifampin Capsules
  Interventions: Drug: SHR2554 and Rifampin

INTERVENTIONS:
Drug: SHR2554 and Rifampin — Single-dose oral administration of SHR2554 and multiple-dose oral administration of Rifampin Capsules

SUMMARY:
The primary objective of the study is to evaluate the effect of Rifampin on pharmacokinetics of healthy Chinese adult subjects after oral administration of SHR2554 tablets. The secondary objective of the study is to evaluate the safety of single-dose oral administration of SHR2554 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent is signed before the trial, and the content, process and possible adverse reactions are fully understood;
2. Be able to complete the study according to the requirements of the test scheme;
3. Healthy male and female subjects aged 18 to 45 years (including both ends) on the date of signing informed consent;
4. The body weight of male subjects is no less than 50 kg and that of female subjects is no less than 45 kg. Body mass index (BMI) is in the range of 19.0-26.0 kg/m2 (including the critical value).

Exclusion Criteria:

1. Participated in blood donation within 3 months before taking the study drug and donate blood ≥400 mL, or received blood transfusion;
2. Allergic constitution, including severe drug allergy or drug allergy history; allergic history of SHR2554 tablets, Rifampin, Rifamycin or their excipients;
3. People who have a history of drug and/or alcohol abuse, have a positive alcohol or drug screening test, or have a history of drug abuse in the past five years or have used drugs within 3 months before the test;
4. Smoking and alcohol addicts (drinking 14 units of alcohol per week: 1 unit = 285 ml beer, 25 ml spirits, or 100 ml wine; smoking ≥ 5 cigarettes a day) and unable to prohibit smoking and alcohol during the test period;
5. Comprehensive physical examination (vital signs, physical examination), routine laboratory examinations (blood routine, blood biochemistry, urine routine, etc.), 12-lead electrocardiogram, chest X-ray, heart color Doppler ultrasound, etc. are abnormal and have clinical significance as judged by the investigator;
6. Echocardiography suggests that the left ventricular ejection fraction (LVEF) is less than 50% or the QT interval (QTcF) corrected by Fridericia method in 12-lead ECG is ≥ 470msec;
7. A clear medical history of primary diseases of important organs such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system, etc., the investigator considers not suitable for participating in this study;
8. Those who have undergone any surgery within 6 months before screening;
9. Hepatotoxic drugs (such as Dapsone, Erythromycin, Fluconazole, Ketoconazole, Rifampin) have been taken for a long period of time (over 7 consecutive days) in the 6 months before screening;
10. Those who have taken any clinical trial drugs within 3 months;
11. Any drug that changes liver enzyme activity was taken within 28 days before taking the study drug;
12. Any prescription or over-the-counter drugs taken within 14 days before taking the study drug;
13. Ingested any vitamin products, health products or Chinese herbal medicine within 14 days before taking the study drug;
14. HCV antibody positive, HIV antibody positive, HBsAg positive, syphilis antibody positive;
15. Ingested grapefruit or products containing grapefruit, food or drink containing caffeine, xanthine or alcohol within 48 hours before taking the study drug; strenuous exercise, or other factors that affect the absorption, distribution, metabolism, and excretion of the study drug;
16. The subjects have a childbearing plan and are unwilling to take effective contraceptive measures 2 weeks before the study administration (only female subjects) and 3 months after the last administration of the drug; those who are fertile and whose serum hCG test is not negative before the study medication;
17. People with a history of fainting needles and blood, have difficulty in blood collection or cannot tolerate venipuncture blood collection;
18. Women during pregnancy and lactation;
19. Subjects with other factors not suitable to participate in this study as considered by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameter: Cmax of SHR2554 | from Day 1 to Day 13
  Peak Plasma Concentration (Cmax) of SHR2554
Pharmacokinetics parameter: AUC of SHR2554 | from Day 1 to Day 13
  Area under the plasma concentration versus time curve (AUC) of SHR2554

SECONDARY OUTCOMES:
Other pharmacokinetics parameter: Tmax of SHR2554 | from Day 1 to Day 13
  Time to maximum plasma concentration (Tmax) of SHR2554
Other pharmacokinetics parameter: T1/2 of SHR2554 | from Day 1 to Day 13
  Half-life of elimination (T1/2) of SHR2554
The incidence and severity of adverse events/serious adverse events | from Day 1 to Day 13
  Based on NCI-CTC AE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu HengRui Medicine Co., Ltd., Shanghai, China

IPD SHARING:
Plan to Share IPD: No